CLINICAL TRIAL: NCT05994339
Title: Radiotherapy Combined With Almonertinib for Stage III EGFR-Mutated Lung Cancer：A Randomized Controlled Clinical Trial
Brief Title: Radiotherapy Combined With Almonertinib for Stage III EGFR-Mutated Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laibin People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Gang, Deputy Director of the Department of Oncology, Laibin People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20220808
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer Stage III
MeSH Terms: conditions — Lung Neoplasms | interventions — aumolertinib; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy Combined with Almonertinib (Experimental): Radiotherapy was administered using Intensity-Modulated Radiation Therapy (IMRT) technique, with a prescribed dose of 60 Gy in 30 fractions. Almonertinib was orally administered at 110 mg per day, starting from the first day of radiotherapy and continued for 42 days until the completion of radiotherapy, followed by continuous medication until disease progression.
  Interventions: Drug: Almonertinib
- Radiotherapy Combined with Chemotherapy (Active Comparator): Radiotherapy was administered using Intensity-Modulated Radiation Therapy (IMRT) technique, with a prescribed dose of 60 Gy in 30 fractions. Chemotherapy with paclitaxel at 135 mg/m2 and cisplatin at 70 mg/m2 was intravenously infused for two cycles during the 1st and 4th weeks. After the completion of radiotherapy, there was a rest period of 4 weeks, followed by continuation of the TP regimen for consolidation chemotherapy for 4 cycles.
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — Radiotherapy was administered using Intensity-Modulated Radiation Therapy (IMRT) technique, with a prescribed dose of 60 Gy in 30 fractions. Almonertinib was orally administered at 110 mg per day, starting from the first day of radiotherapy and continued for 42 days until the completion of radiotherapy, followed by continuous medication until disease progression.
  Other Names: Intensity-Modulated Radiation Therapy(IMRT)

SUMMARY:
Study Object: Stage III lung cancer with epidermal growth factor receptor (EGFR) sensitive mutation.

Study Method: The study subjects will be randomly assigned to the intervention group and the control group. The intervention group will receive radiotherapy combined with erlotinib treatment, while the control group will receive concurrent radiotherapy combined with chemotherapy. The differences in short-term efficacy, long-term efficacy, and incidence of adverse reactions between the two groups will be observed.

Observation Indicators: Short-term efficacy indicators: Complete remission (CR) rate, partial remission (PR) rate, and objective response rate (ORR). Long-term efficacy indicators: Overall survival (OS) and progression-free survival (PFS). Adverse reaction indicators: Incidence of lung toxicity, hematological toxicity, and gastrointestinal reactions.

DETAILED DESCRIPTION:
The following tasks need to be completed at the time of enrollment: screening, signing the informed consent form, random assignment according to the randomization table, detailed patient medical history, physical examination, and collection of baseline chest-enhanced CT as imaging data before treatment.

All eligible patients who meet the baseline inclusion criteria will be enrolled using an online central randomization system, with the following stratification factors: disease staging at the beginning of the study treatment (ⅢA vs ⅢB vs ⅢC), histology (adenocarcinoma vs. others), and EGFR mutation status (exon 19 vs. exon 21). Patients will be randomly assigned in a 1:1 ratio.

In the intervention group，Radiotherapy was administered using Intensity-Modulated Radiation Therapy (IMRT) technique, with a prescribed dose of 60 Gy in 30 fractions. Ametinib was orally administered at 110 mg per day, starting from the first day of radiotherapy and continued for 42 days until the completion of radiotherapy, followed by continuous medication until disease progression. In the control group，Radiotherapy was administered using Intensity-Modulated Radiation Therapy (IMRT) technique, with a prescribed dose of 60 Gy in 30 fractions. Chemotherapy with paclitaxel at 135 mg/m2 and cisplatin at 70 mg/m2 was intravenously infused for two cycles during the 1st and 4th weeks. After the completion of radiotherapy, there was a rest period of 4 weeks, followed by continuation of the TP regimen for consolidation chemotherapy for 4 cycles.

Follow-up will take place from August 30, 2023, to December 30, 2025, based on the time of death. Chest and upper abdominal enhanced CT, cervical supraclavicular lymph node color Doppler ultrasound, head MRI, whole-body bone scan, and other examinations will be performed at treatment completion, 1 month after treatment completion, 3 months after treatment completion, every 3 months within 2 years, and every 6 months in the 3rd year for efficacy and survival evaluation.

Statistical Analysis:

① Stratified (based on disease stage at the beginning of the study treatment, histology, and EGFR mutation status) and unstratified log-rank tests will be used to compare Progression-Free Survival (PFS) and Overall Survival (OS) at a two-sided significance level of 0.05. The median PFS and corresponding 95% confidence intervals (CI) for both groups will be calculated.

② Cox proportional hazards models will be used to estimate Hazard Ratios (HRs) and 95% CI for PFS and OS. PFS and OS curves will be estimated using the Kaplan-Meier method.

③ Fisher's exact test will be used to compare the difference in Objective Response Rate (ORR) between the two groups. The difference in ORR and its 95% CI will be presented together using the normal approximation method.

ELIGIBILITY:
Inclusion Criteria:

* Patients initially diagnosed with lung cancer through imaging and pathological examination.

  * Genetic testing confirms EGFR-sensitive mutations.

    * Staging according to the international eighth edition of lung cancer TNM is between stage ⅢA to ⅢC.

      * Age between 18 to 80 years old, without severe organ diseases such as heart, liver, kidney, etc.

        ⑤ General condition assessed with a performance status (PS) score of ≤2 points.

Exclusion Criteria:

* ① Patients with upper gastrointestinal physiological disorders, malabsorption syndrome, intolerance to oral medications, or peptic ulcers.

  * Patients who have received previous radiotherapy or chemotherapy for lung conditions.

    * Patients with concomitant chronic obstructive pulmonary disease, atelectasis, or other conditions that cause difficulties in lesion measurements.

      * Patients with active pulmonary tuberculosis. ⑤ Patients with respiratory failure. ⑥ Patients with allergies to the investigational drugs used in this study. ⑦ Pregnant or lactating women. ⑧ Patients with any other diseases, neurological or metabolic disorders, physical examination or laboratory findings that may raise reasonable suspicions of certain diseases or conditions, which would either disqualify the use of the investigational drugs or place the subjects at high risk of treatment-related complications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
overall survival(OS) | 2 years
  the duration from treatment initiation to mortality resulting from any reason.

SECONDARY OUTCOMES:
progression-free survival (PFS) | 2 years
  the period from treatment initiation to the first documented progressive disease (PD) or death.
Objective Response Rate (ORR): | 3 months
  Complete Remission (CR) is defined as complete disappearance of lesions and maintained for more than 1 month; Partial Remission (PR) is defined as more than 50% reduction in lesion volume and maintained for more than 1 month; Effective rate (ORR) is calculated as CR + PR.

IPD SHARING:
Plan to Share IPD: No